CLINICAL TRIAL: NCT01186094
Title: Percutaneous Treatment of LONG Native Coronary Lesions With Drug-Eluting Stent-IV: Sirolimus vs. Zotarolimus-eluting Stent
Brief Title: Percutaneous Treatment of LONG Native Coronary Lesions With Drug-Eluting Stent-IV: (LONG-DES-IV)
Acronym: LONG-DES-IV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other); Medtronic (Industry)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, MD,PhD, Chairman,Heart Institute, Asan Medical Center,University of Ulsan,College of Medicine, CardioVascular Research Foundation, Korea
Organization: CardioVascular Research Foundation, Korea (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2008-0086
Record Dates: First submitted 2009-10-18; First posted 2010-08-23 (Estimated); Last update posted 2012-08-08 (Estimated); Status verified 2012-08

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Stent
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cypher (Active Comparator): Sirolimus-eluting stent
  Interventions: Device: Cypher
- Endeavor Resolute (Active Comparator): Zotarolimus-eluting Stent
  Interventions: Device: Endeavor Resolute

INTERVENTIONS:
Device: Cypher — Sirolimus-eluting stent
  Other Names: Sirolimus-eluting stent
  Arms: Cypher
Device: Endeavor Resolute — Zotarolimus-eluting Stent
  Other Names: Zotarolimus-eluting Stent
  Arms: Endeavor Resolute

SUMMARY:
This randomized study is a multi-center, randomized, study to compare the efficacy of sirolimus (Cypher) versus zotarolimus-eluting stent (Endeavor Resolute) implantation for long coronary lesions.

DETAILED DESCRIPTION:
Following angiography, patients with significant diameter stenosis >50% and lesion length (> 25mm) requiring single or multiple long-stent placement (total stent length>28mm) by visual estimation and eligible for LONG-DES IV trial inclusion and exclusion criteria will be randomized 1:1 to a) CYPHER and b) ENDEAVOR RESOLUTE stent by the stratified randomization method.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be at least 18 years of age.
* Significant native coronary artery stenosis (>50% by visual estimate) with lesion length of more than 25mm, which requiring single or multiple long stent placement (>=28mm)
* Patients with silent ischemia, stable or unstable angina pectoris, ad Non-ST-elevation myocardial infarction
* The patient or guardian agrees to the study protocol and the schedule of clinical and angiographic follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethical Committee of the respective clinical site.

Exclusion Criteria:

* Any contraindication to any of the following medications: aspirin, heparin, clopidogrel, stainless steel, contrast agents, sirolimus, or everolimus.
* An elective surgical procedure is planned that would necessitate interruption of antiplatelet drugs during the first 6 months post enrollment.
* Acute ST-segment-elevation MI or cardiogenic shock
* Terminal illness with life expectancy <1 year
* Patients who are actively participating in another drug or device investigational study, which have not completed the primary endpoint follow-up period.
* In-stent restenosis at target vessel (either bare metal stent or drug-eluting stent segment, non-target vessel ISR is permitted)
* Patients with EF<30%.
* Serum creatinine level >=3.0mg/dL or dependence on dialysis.
* Patients with left main stem stenosis (>50% by visual estimate).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 502 (Actual)
Dates: Start 2009-05; Primary Completion 2011-04 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
In-segment late luminal loss | 9 month follow-up

SECONDARY OUTCOMES:
All Death | 1 year
Cardiac death | 1 year
Myocardial infarction (MI) | 1 year
Composite of death or MI | 1 year
Composite of cardiac death or MI | 1 year
Target vessel revascularization (ischemia-driven and clinically-driven) | 1 year
Target lesion revascularization (ischemia-driven and clinically-driven) | 1 year
Target-vessel failure (death from any cause, myocardial infarction, and ischemic-driven target-vessel revascularization) | 12 months
Stent thrombosis (ARC criteria) | 1 year
In-stent late loss at 9 month angiographic follow-up | at 9 month angiographic follow-up
In-stent and in-segment restenosis at 9 month angiographic follow-up | at 9 month angiographic follow-up
Angiographic pattern of restenosis at 9 month angiographic follow-up | at 9 month angiographic follow-up
Volume of intimal hyperplasia at 9 month IVUS follow-up (sub-study) | at 9 month angiographic follow-up
Incidence of late stent malapposition at 9 month IVUS follow-up (sub-study) | at 9 month angiographic follow-up
Procedural success defined as achievement of a final diameter stenosis of <30% by QCA using any percutaneous method, without the occurrence of death, Q wave MI, or repeat revascularization of the target lesion during the hospital stay. | at 3 days in average
  At discharge from the index hospitalization (normal hospitalization is from 3 -4 days.)
All death | one month
All death | 9 months
Cardiac death | one month
Cardiac death | 9 months
Myocardial infarction (MI) | one month
Myocardial infarction (MI) | 9 months
Composite of death or MI | one month
Composite of death or MI | 9 months
Composite of cardiac death or MI | one month
Composite of cardiac death or MI | 9 months
Target vessel revascularization (ischemia-driven and clinically-driven) | one month
Target vessel revascularization (ischemia-driven and clinically-driven) | 9 months
Target lesion revascularization (ischemia-driven and clinically-driven) | one month
Target lesion revascularization (ischemia-driven and clinically-driven) | 9 months
Stent thrombosis (ARC criteria) | one month
Stent thrombosis (ARC criteria) | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Jung Park, MD, PhD, Principal Investigator — Department of Medicine, Asan Medical Center, University of Ulsan College of Medicine
Locations (12):
- South Korea (12):
  - Stcarollo Hospital, Suncheon, Cheon-nam
  - Konyang University Hospital, Daejeon, Chungcheongnam-do
  - Wonju Christian Hospital, Wŏnju, Gangwon-do
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si, Gyeonggi-do
  - Inje University Ilsan Paik Hospital, Ilsan, Gyeonggi-do
  - Yeungnam University Medical Center, Daegu, Kyung-book
  - Busan Paik Hospital, Busan
  - Dong-A University Medical Center, Busan
  - Soonchunhyang University Cheonan Hospital, Cheonan
  - Gangwon National University Hospital, Chuncheon
  - Asan Medical Center, Seoul
  - Kyung Hee University Medical Hospital, Seoul

REFERENCES:
- [Derived] Ahn JM, Park DW, Kim YH, Song H, Cho YR, Kim WJ, Lee JY, Kang SJ, Lee SW, Lee CW, Park SW, Yun SC, Han S, Lee SY, Lee BK, Cho JH, Yang TH, Lee NH, Yang JY, Park JS, Shin WY, Kim MH, Bae JH, Kim MK, Yoon J, Park SJ. Comparison of resolute zotarolimus-eluting stents and sirolimus-eluting stents in patients with de novo long coronary artery lesions: a randomized LONG-DES IV trial. Circ Cardiovasc Interv. 2012 Oct;5(5):633-40. doi: 10.1161/CIRCINTERVENTIONS.111.965673. Epub 2012 Oct 9. PMID 23048051